CLINICAL TRIAL: NCT00646360
Title: Effects of Prenatal DHA Supplements on Infant Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Instituto Nacional de Salud Publica, Mexico (Other); Instituto Mexicano del Seguro Social (Other Government); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Usha Ramakrishnan, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00024976; 5R01HD043099 (NIH); 5R03HD087606 (NIH)
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Pregnancy
Keywords: birth size, gestational age, development, child growth,; prenatal nutrition, DHA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHA arm (Experimental): Docosahexonic acid (DHA) (400 mg/day). Pregnant women attending the IMSS General Hospital I are recruited between 18-22 wks gestation and assigned randomly to receive either DHA (400 mg) or a placebo daily until delivery.
  Interventions: Dietary Supplement: DHA
- Placebo arm (Placebo Comparator): Pregnant women attending the IMSS General Hospital I are recruited between 18-22 wks gestation and assigned randomly to receive either DHA (400 mg) or a placebo daily until delivery.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: DHA — 400 mg/d of docosahexanoic acid (DHA) during pregnancy
  Other Names: Martek Algal DHA
  Arms: DHA arm
Dietary Supplement: Placebo — 2 tablets daily during pregnancy
  Other Names: Specially formulated by Martek Biosciences
  Arms: Placebo arm

SUMMARY:
This research study research is about the significance of polyunsaturated fatty acids (PUFAs) for human development. Specifically, the study team will assess the effect of docosahexanoic acid (DHA) supplementation during pregnancy on infant growth and development through a randomized controlled intervention trial in Cuernavaca, Mexico. This is a collaborative effort between the Rollins School of Public Health, Emory University, the Instituto Nacional de Salud Publica (INSP) and the Instituto Mexicano del Seguro Social (IMSS), Cuernavaca, Mexico. Pregnant women attending the IMSS General Hospital I are recruited between 18-22 weeks gestation and assigned randomly to receive either DHA (400 mg) or a placebo daily until delivery. The main study outcomes include a) birth outcomes: birth size, gestational age, cord blood levels of DHA and neurodevelopment b) maternal blood and breast milk DHA levels at 1 and 3 months post-partum, c) postnatal growth and development during the first 5 years of age and d) infant DHA status at 3, 12 and 18 months.

DETAILED DESCRIPTION:
This research study is about the significance of polyunsaturated fatty acids (PUFAs) for human development. Specifically, the study team will assess the effect of docosahexanoic acid (DHA) supplementation during pregnancy on infant growth and development through a randomized controlled intervention trial in Cuernavaca, Mexico. This is a collaborative effort between the Rollins School of Public Health, Emory University, the Instituto Nacional de Salud Publica (INSP) and the Instituto Mexicano del Seguro Social (IMSS), Cuernavaca, Mexico. Pregnant women attending the IMSS General Hospital I are recruited between 18-22 wks gestation and assigned randomly to receive either DHA (400 mg) or a placebo daily until delivery. The main study outcomes include a) birth outcomes: birth size, gestational age, cord blood levels of DHA and neurodevelopment b) maternal blood and breast milk DHA levels at 1 and 3 mo post-partum c) postnatal growth and development during the first 5 years of age and d) infant DHA status at 3, 12 and 18 mo. All data collection is carried out at the study headquarters (IMSS) except for home environment that is assessed during home visits. Physical growth (length, weight, and head circumference) and infant and child development (visual and auditory evoked potentials, visual attention, Bayley scales of infant development, McCarthy child development score, Hearts and Flowers stroop test, and other computerized child development tests) are measured at birth, 1, 3, 6, 9, 12, 18, 24, 36 months and at 4 and 5 years of age by trained workers. Data are also obtained on socioeconomic status, obstetric history, maternal diet, anthropometry and intelligence, quality of home environment and infant feeding practices. Data analysis will include group comparisons (intent-to-treat) after ensuring effectiveness of randomization, and structural equation modeling to examine the various pathways by which DHA supplementation during pregnancy affects child growth and development. The findings of this project will contribute significantly to our understanding of the functional consequences of DHA supplementation during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* 18-22 weeks pregnant (based on last menstrual period)
* 18 - 35 years old
* Resident of Cuernavaca who intends to deliver at the IMSS General Hospital I and remain in the area for the 2 years following recruitment
* Intends to predominantly breastfeed infant until 3 months of age
* Agrees to participate with informed consent

Exclusion criteria

* High risk pregnancy: If documented in the clinical record at recruitment and will include history and prevalence of abruptio placentae, any serious bleeding episode in the current pregnancy, gestational diabetes, pregnancy induced hypertension, maternal toxoplasmosis infection during pregnancy, coagulation disorders, thrombocytopenia or chronic vascular, renal or systemic disease and drug use.
* Lipid metabolism (hyperlipidemia) and/or absorption disorders
* Regular intake of fish oil or DHA supplements during pregnancy
* Chronic use of medication for illnesses like epilepsy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1094 (Actual)
Dates: Start 2005-02 (Actual); Primary Completion 2013-01-03 (Actual); Study Completion 2014-08-16 (Actual)

PRIMARY OUTCOMES:
Birth size | Birth
  Birth size will be determined by measuring the newborn, a baby's length is measured from the top of their head to the bottom of one of their heels.
Gestational age | Birth
  Gestational age is measured in weeks, from the first day of the woman's last menstrual cycle to the current date.
Changes in visual evoked potentials | 3 and 6 months of age
  Visual evoked potential (VEP) is an electrical signal emanated from the brain while a visual stimulus is presented to the subject in a time locked manner. The VEP can be used as a diagnostic tool to detect ocular diseases in patients with visually impaired. VEP response can also be used to detect eye diseases like glaucoma, diabetic retinopathy, multiple sclerosis, ocular hypertension, loss of peripheral (side) vision, macular degeneration and color blindness.
Changes in infant weight | Birth, months 1, 3, 6, 9, 12, 18, 24, 36 and at 4 and 5 years of age
  Infant weight is measured in kilograms (kg) and weight is measured in the hospital and at all check-ups.
Changes in infant height | Birth, months 1, 3, 6, 9, 12, 18, 24, 36 and at 4 and 5 years of age
  Infants will be measured in the hospital and at all check-ups. Height is measured in centimeters (cm).
Changes In infant head circumference | Birth, months 1, 3, 6, 9, 12, 18, 24, 36 and at 4 and 5 years of age
  Head circumference or OFC [occipital frontal circumference] is measured over the most prominent part on the back of the head (occiput) and just above the eyebrows (supraorbital ridges). This can be translated to mean the largest circumference of the head. Head circumference is measured in centimeters (cm).
Changes in auditory evoked potentials | 1 and 3 months of age
  A brainstem auditory evoked response (BAER) test measures how the brain processes the sounds a person hears. The BAER test records the subject's brainwaves in response to clicks or other audio tones that are played for them.
Changes in child development score | 1, 1.5 and 5 years of age
  The Bayley Scales of Infant Development -II are used to assess child development during the first two years of life while The McCarthy Scales of Children's Abilities (MSCA) is a psychological instrument for young children that measures cognitive ability in six domain areas: Verbal, Perceptual-Performance, Quantitative, General Cognitive, Memory, and Motor at age 5 y.
Changes in Hearts and Flowers Stroop Test | 5 years of age
  This tests working memory, response inhibition, and task switching/cognitive flexibility . The task requires participants to press a response button that is either on the same side (congruent) or opposite side (incongruent) of an image. When children see an image of a heart, they are instructed to press the corresponding directional arrow button on a keyboard. When children see an image of a flower, they are instructed to press the opposite directional arrow button on the keyboard . The task consists of three separate levels that contain only congruent trials (12 trials total), only incongruent trials (12 trials total), and mixed congruent and incongruent trials respectively (33 trials total). Images are presented on a computer monitor. Before both the congruent and incongruent trial blocks, a training period is administered which consists of 5 trials. The child is unable to advance to the next question until they respond correctly.

SECONDARY OUTCOMES:
Changes Immune function | first 6 months of life
Changes in Morbidity | Birth, months 1, 3, 6, 9, 12, 18, 24, 36 and at 4 and 5 years of age
  Changes in morbidity (health) factors will be assessed.
Cognitive outcomes at age 7 years of age | At 7 year follow up
  The cognitive intelligence test WAIS-IV offers compound scores that reflect the intellectual functioning of 4 cognitive areas (verbal understanding, perceptive reasoning, working memory and processing speed). It also offers a compound score that reflects intellectual aptitude in general (Intelligence quotient).

CONTACTS AND LOCATIONS:
Overall Officials: Usha Ramakrishnan, Ph.D., Principal Investigator — Emory University
Locations (1):
- IMSS General Hospital I, Cuernavaca, Morelos, Mexico

REFERENCES:
- [Derived] Wimalasena ST, Ramirez-Silva CI, Gonzalez Casanova I, Stein AD, Sun YV, Rivera JA, Demmelmair H, Koletzko B, Ramakrishnan U. Effects of prenatal docosahexaenoic acid supplementation on offspring cardiometabolic health at 11 years differs by maternal single nucleotide polymorphism rs174602: follow-up of a randomized controlled trial in Mexico. Am J Clin Nutr. 2023 Dec;118(6):1123-1132. doi: 10.1016/j.ajcnut.2023.10.005. Epub 2023 Oct 14. PMID 37839707
- [Derived] Gonzalez Casanova I, Schoen M, Tandon S, Stein AD, Barraza Villarreal A, DiGirolamo AM, Demmelmair H, Ramirez Silva I, Feregrino RG, Rzehak P, Stevenson I, Standl M, Schnaas L, Romieu I, Koletzko B, Ramakrishnan U. Maternal FADS2 single nucleotide polymorphism modified the impact of prenatal docosahexaenoic acid (DHA) supplementation on child neurodevelopment at 5 years: Follow-up of a randomized clinical trial. Clin Nutr. 2021 Oct;40(10):5339-5345. doi: 10.1016/j.clnu.2021.08.026. Epub 2021 Sep 11. PMID 34543890
- [Derived] Tandon S, Gonzalez-Casanova I, Barraza-Villarreal A, Romieu I, Demmelmair H, Jones DP, Koletzko B, Stein AD, Ramakrishnan U. Infant Metabolome in Relation to Prenatal DHA Supplementation and Maternal Single-Nucleotide Polymorphism rs174602: Secondary Analysis of a Randomized Controlled Trial in Mexico. J Nutr. 2021 Nov 2;151(11):3339-3349. doi: 10.1093/jn/nxab276. PMID 34494106
- [Derived] Barrios PL, Garcia-Feregrino R, Rivera JA, Barraza-Villarreal A, Hernandez-Cadena L, Romieu I, Gonzalez-Casanova I, Ramakrishnan U, Hoffman DJ. Height Trajectory During Early Childhood Is Inversely Associated with Fat Mass in Later Childhood in Mexican Boys. J Nutr. 2019 Nov 1;149(11):2011-2019. doi: 10.1093/jn/nxz157. PMID 31334762
- [Derived] Gonzalez-Casanova I, Stein AD, Barraza-Villarreal A, Feregrino RG, DiGirolamo A, Hernandez-Cadena L, Rivera JA, Romieu I, Ramakrishnan U. Prenatal exposure to environmental pollutants and child development trajectories through 7 years. Int J Hyg Environ Health. 2018 May;221(4):616-622. doi: 10.1016/j.ijheh.2018.04.004. Epub 2018 Apr 22. PMID 29699913
- [Derived] Gutierrez-Delgado RI, Barraza-Villarreal A, Escamilla-Nunez C, Hernandez-Cadena L, Garcia-Feregrino R, Shackleton C, Ramakrishnan U, Sly PD, Romieu I. Effect of omega-3 fatty acids supplementation during pregnancy on lung function in preschoolers: a clinical trial. J Asthma. 2019 Mar;56(3):296-302. doi: 10.1080/02770903.2018.1452934. Epub 2018 Apr 4. PMID 29617210
- [Derived] Gutierrez-Gomez Y, Stein AD, Ramakrishnan U, Barraza-Villarreal A, Moreno-Macias H, Aguilar-Salinas C, Romieu I, Rivera JA. Prenatal Docosahexaenoic Acid Supplementation Does Not Affect Nonfasting Serum Lipid and Glucose Concentrations of Offspring at 4 Years of Age in a Follow-Up of a Randomized Controlled Clinical Trial in Mexico. J Nutr. 2017 Feb;147(2):242-247. doi: 10.3945/jn.116.238329. Epub 2016 Dec 21. PMID 28003539
- [Derived] Ramakrishnan U, Gonzalez-Casanova I, Schnaas L, DiGirolamo A, Quezada AD, Pallo BC, Hao W, Neufeld LM, Rivera JA, Stein AD, Martorell R. Prenatal supplementation with DHA improves attention at 5 y of age: a randomized controlled trial. Am J Clin Nutr. 2016 Oct;104(4):1075-1082. doi: 10.3945/ajcn.114.101071. Epub 2016 Sep 7. PMID 27604770
- [Derived] Gonzalez-Casanova I, Rzehak P, Stein AD, Garcia Feregrino R, Rivera Dommarco JA, Barraza-Villarreal A, Demmelmair H, Romieu I, Villalpando S, Martorell R, Koletzko B, Ramakrishnan U. Maternal single nucleotide polymorphisms in the fatty acid desaturase 1 and 2 coding regions modify the impact of prenatal supplementation with DHA on birth weight. Am J Clin Nutr. 2016 Apr;103(4):1171-8. doi: 10.3945/ajcn.115.121244. Epub 2016 Feb 24. PMID 26912491
- [Derived] Ramakrishnan U, Stinger A, DiGirolamo AM, Martorell R, Neufeld LM, Rivera JA, Schnaas L, Stein AD, Wang M. Prenatal Docosahexaenoic Acid Supplementation and Offspring Development at 18 Months: Randomized Controlled Trial. PLoS One. 2015 Aug 11;10(8):e0120065. doi: 10.1371/journal.pone.0120065. eCollection 2015. PMID 26262896
- [Derived] Gonzalez-Casanova I, Stein AD, Hao W, Garcia-Feregrino R, Barraza-Villarreal A, Romieu I, Rivera JA, Martorell R, Ramakrishnan U. Prenatal Supplementation with Docosahexaenoic Acid Has No Effect on Growth through 60 Months of Age. J Nutr. 2015 Jun;145(6):1330-4. doi: 10.3945/jn.114.203570. Epub 2015 Apr 29. PMID 25926416
- [Derived] Escamilla-Nunez MC, Barraza-Villarreal A, Hernandez-Cadena L, Navarro-Olivos E, Sly PD, Romieu I. Omega-3 fatty acid supplementation during pregnancy and respiratory symptoms in children. Chest. 2014 Aug;146(2):373-382. doi: 10.1378/chest.13-1432. PMID 24626819
- [Derived] Hernandez E, Barraza-Villarreal A, Escamilla-Nunez MC, Hernandez-Cadena L, Sly PD, Neufeld LM, Ramakishnan U, Romieu I. Prenatal determinants of cord blood total immunoglobulin E levels in Mexican newborns. Allergy Asthma Proc. 2013 Sep-Oct;34(5):e27-34. doi: 10.2500/aap.2013.34.3688. PMID 23998234
- [Derived] Stein AD, Wang M, Rivera JA, Martorell R, Ramakrishnan U. Auditory- and visual-evoked potentials in Mexican infants are not affected by maternal supplementation with 400 mg/d docosahexaenoic acid in the second half of pregnancy. J Nutr. 2012 Aug;142(8):1577-81. doi: 10.3945/jn.112.162461. Epub 2012 Jun 27. PMID 22739364
- [Derived] Imhoff-Kunsch B, Stein AD, Martorell R, Parra-Cabrera S, Romieu I, Ramakrishnan U. Prenatal docosahexaenoic acid supplementation and infant morbidity: randomized controlled trial. Pediatrics. 2011 Sep;128(3):e505-12. doi: 10.1542/peds.2010-1386. Epub 2011 Aug 1. PMID 21807696
- [Derived] Stein AD, Wang M, Martorell R, Neufeld LM, Flores-Ayala R, Rivera JA, Ramakrishnan U. Growth to age 18 months following prenatal supplementation with docosahexaenoic acid differs by maternal gravidity in Mexico. J Nutr. 2011 Feb;141(2):316-20. doi: 10.3945/jn.110.128215. Epub 2010 Dec 22. PMID 21178082
- [Derived] Imhoff-Kunsch B, Stein AD, Villalpando S, Martorell R, Ramakrishnan U. Docosahexaenoic acid supplementation from mid-pregnancy to parturition influenced breast milk fatty acid concentrations at 1 month postpartum in Mexican women. J Nutr. 2011 Feb;141(2):321-6. doi: 10.3945/jn.110.126870. Epub 2010 Dec 22. PMID 21178076
- [Derived] Ramakrishnan U, Stein AD, Parra-Cabrera S, Wang M, Imhoff-Kunsch B, Juarez-Marquez S, Rivera J, Martorell R. Effects of docosahexaenoic acid supplementation during pregnancy on gestational age and size at birth: randomized, double-blind, placebo-controlled trial in Mexico. Food Nutr Bull. 2010 Jun;31(2 Suppl):S108-16. doi: 10.1177/15648265100312S203. PMID 20715595